CLINICAL TRIAL: NCT02235298
Title: Effects of Dapagliflozin on Epicardial Fat in Subjects With Type 2 Diabetes
Brief Title: Dapagliflozin Effects on Epicardial Fat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20140671
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes
Keywords: epicardial fat; diabetes; dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin and Metformin Group (Experimental): Participants in this group will receive Dapagliflozin in addition to Metformin for 6 months.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Metformin and Placebo Group (Active Comparator): Participants in this group will receive Metformin and Placebo for 6 months.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 5 mg taken orally once daily. After 2 weeks, if there are no safety issues as per treating physician discretion, the dose can be titrated up to 10 mg orally taken once daily.
  Other Names: Farxiga
  Arms: Dapagliflozin and Metformin Group
Drug: Metformin — 500 mg taken orally twice daily to a maximum of 1000 mg twice daily to achieve a fasting glucose between 80-140 md/dL
Drug: Placebo — Placebo pill taken once daily to mimic Dapagliflozin
  Arms: Metformin and Placebo Group

SUMMARY:
The purpose of this research study is to learn about the effect of Dapagliflozin (Farxiga) on the fat of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, as defined by ADA criteria
* HbA1c < 8% measured at least 1 week prior to the study
* BMI ≥27 kg/m2
* Pre-treatment with Metformin as monotherapy
* Age > 18 and < 65 years old
* Normal and stable hemodynamic status

Exclusion Criteria:

* Known contra-indications to Farxiga, in accordance with risks and safety information included in the latest updated Prescribing Information
* Type 1 diabetes, as defined by American Diabetes Association (ADA) criteria
* Insulin dependent or treated type 2 diabetes
* Current use of other SGLT2 inhibitors, Glucagon Like Peptide -1 (GLP- 1) analogs or Dipeptidyl Peptidase 4 (DPP4) inhibitors
* Glomerular Filtration Rate (GFR) < 60 mL/min/1.73 m2
* Signs or symptoms of hypovolemia
* Patients with poor glycemic control (HbA1c ≥ 8%) will be excluded to maximize long-term patient retention without need
* History of diabetes ketoacidosis
* Patients with active bladder cancer or with a prior history of bladder cancer
* Acute or chronic infective, including genital mycotic infections
* Clinical signs or symptoms of New York Heart Association (NYHA) class III-IV heart failure
* Clinical or laboratory evidences of chronic active liver diseases
* Acute or chronic infective diseases
* Cancer or chemotherapy
* Current use of systemic corticosteroids or in the 3 months prior this study
* Known or suspected allergy to Dapagliflozin, excipients, or related products
* Pregnant, breast-feeding or the intention of becoming pregnant
* Females of childbearing potential who are not using adequate contraceptive methods

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Iacobellis, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin and Metformin Group | Metformin and Placebo Group
Started | 50 | 50
Completed | 42 | 42
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 6 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin and Metformin Group | Metformin and Placebo Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9) | 51 (11) | 51.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 47
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Epicardial Fat Thickness
Description: Epicardial fat thickness will be measured in millimeters by treating physician using echocardiography at Baseline, 12 weeks, 24 weeks
Time Frame: At Baseline, 12 weeks, 24 weeks
Population: Data is reported only for the participants that completed the study intervention.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dapagliflozin and Metformin Group | Metformin and Placebo Group
Number analyzed (Participants) | 42 | 42
mm
  Baseline | 8.6 (2.2) | 8.0 (2.5)
  12 Weeks | 7.2 (2.3) | 7.4 (2.5)
  24 Weeks | 6.7 (2.1) | 7.5 (2.4)

2. Secondary Outcome: Left Ventricular Mass (LVM)
Description: LVM will be measured in g/m^2 by treating physician using echocardiography at baseline, Week 12 and Week 24
Time Frame: At Baseline, Week 12 and Week 24
Population: Due to time and technical limitations, LVM data were not collected for all participants that completed the study intervention.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Dapagliflozin and Metformin Group | Metformin and Placebo Group
Number analyzed (Participants) | 33 | 24
g/m^2
  Baseline | 129 (13) | 130 (19)
  Week 12 | 127 (18) | 128 (20)
  Week 24 | 122 (19) | 122 (20)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Dapagliflozin and Metformin Group | Metformin and Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 8/50 | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin and Metformin Group (N=50) | Metformin and Placebo Group (N=50)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Balanitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 2 (2)
Frequency of Urination (Renal and urinary disorders) | 6 (6) | 0 (0)
Dysuria (Renal and urinary disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT02235298/Prot_SAP_000.pdf